CLINICAL TRIAL: NCT02527304
Title: Adaptive Staged Stereotactic Body Radiation Therapy in Treating Patients With Spinal Metastases That Cannot Be Removed by Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-4957; NCI-2015-01222 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 007683; 2015-4957 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Melanoma; Metastatic Malignant Neoplasm in the Spine; Renal Cell Carcinoma; Soft Tissue Sarcoma; Spinal Cord Compression
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Sarcoma; Spinal Cord Compression | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment (adaptive staged SBRT) (Experimental): Patients undergo adaptive staged SBRT. Within 14-21 days, patients may undergo a second treatment of adaptive staged SBRT at the discretion of the treating physician based on clinical parameters, diagnostic interval imaging, and achievement of spinal cord dose constraints.
  Interventions: Radiation: Image-Guided Adaptive Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Image-Guided Adaptive Radiation Therapy — Undergo adaptive staged SBRT
  Other Names: IGART
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo adaptive staged SBRT
  Other Names: SBRT

SUMMARY:
This pilot clinical trial studies adaptive staged stereotactic body radiation therapy (SBRT) in treating patients with spinal metastases that cannot be removed by surgery. SBRT is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue. Adaptive SBRT uses information gathered during treatment to inform, guide, and alter future radiation treatments. Staged SBRT uses multiple treatments separated by 2-3 weeks. Giving adaptive staged SBRT may work better in treating spinal metastases that cannot be removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of single-fraction radiotherapy to provide a short-interval treatment response in patients with metastatic epidural spinal cord compression (MESCC), such that additional stereotactic radiotherapy to full therapeutic doses can be delivered while respecting spinal cord constraints, based on the following metrics: shortest distance between gross disease and the spinal cord before and after treatment; epidural tumor volume before and after treatment; and extent of epidural compression before and after treatment.

SECONDARY OBJECTIVES:

I. To evaluate pain control using the Numerical Rating Pain Scale (NRPS) before and after treatment.

II. To evaluate patient quality of life using the Functional Assessment of Cancer Therapy-General (FACT-G) before and after treatment.

III. To evaluate functional outcomes using ambulation score and standardized neurologic exams before and after treatment.

OUTLINE:

Patients undergo adaptive staged SBRT. Within 14-21 days, patients may undergo a second treatment of adaptive staged SBRT at the discretion of the treating physician based on clinical parameters, diagnostic interval imaging, and achievement of spinal cord dose constraints.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Localized spine metastasis from the cervical (C)1 to lumbar (L)5 levels with documented epidural cord compression by a screening imaging study (magnetic resonance imaging [MRI] or computed tomography [CT] myelogram); site may have a maximal involvement of 2 contiguous vertebral bodies; patients with other visceral metastasis, and radioresistant tumors (including soft tissue sarcomas, melanomas, and renal cell carcinomas) are eligible
* History/physical examination by the treating physician within 24 hours prior to registration
* Neurological and functional examination within 24 hours prior to registration by the treating physician
* Negative serum pregnancy test
* MRI (contrast is not required but strongly recommended) or CT myelogram of the involved spine within 1 week prior to registration to determine the extent of the spine involvement
* Numerical rating pain scale within 1 week prior to registration; documentation of the patient's initial pain score is required; patients taking medication for pain at the time of registration are eligible
* Women of childbearing potential must:

  * Have a negative serum or urine pregnancy test within 72 hours prior to the start of study therapy
  * Agree to utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study therapy is completed
  * Be advised of the importance of avoiding pregnancy during trial participation and the potential risks of an unintentional pregnancy
* All patients must sign study specific informed consent prior to study entry or within 1 week of first treatment, provided other criteria were met
* Patients considered for enrollment are strongly recommended to have been discussed at multidisciplinary tumor board with input from surgery, medical oncology and radiation oncology prior to enrollment

Exclusion Criteria:

* Histologies of myeloma or lymphoma
* Cord compression at 2 non-contiguous sites in the spine
* Favorable candidates for surgical decompression by prior documented criteria
* Spine instability as determined by Spinal Instability Neoplastic Score (SINS) score > 12
* > 50% loss of vertebral body height
* Bony retropulsion causing neurologic abnormality
* Prior radiation to the index spine
* Patients who cannot obtain a contrast-enhanced MRI or CT myelogram due to allergy, renal failure or other medical contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhur Garg, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Adaptive Staged SBRT)
Started | 24
Completed | 12
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: total patients enrolled
Arm/Group | Treatment (Adaptive Staged SBRT)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 14
Age, Continuous [Mean (Full Range); unit: years] | 66.5 [32 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 4
  More than one race | 5
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24
Numeric Pain Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. 0 indicates "no pain", and 10 indicates "worst possible pain."
  units on a scale | 4.31 (3)

OUTCOME MEASURES:

1. Primary Outcome: Distance Between the Gross Disease and Spinal Cord (Cord-disease Distance, CDD) of at Least 3mm After Treatment.
Description: Cord-disease distance of at least 3mm in shortest axial distance after treatment. Data was summarized using standard descriptive statistics; formal hypothesis testing was not performed. Confidence intervals for the true proportion were computed using Clopper-Pearson exact confidence interval were not conducted. Since this was a feasibility, study no power calculation was done.
Time Frame: Up to 10 weeks after first treatment
Population: Data was not collected and analyzed for 9 participants due to no post-treatment imaging being obtained. Imaging was unable to be conducted for these participants due to either a decline in subjects' clinical status or death. Confidence intervals were not determined given data limitations and had no impact due to feasibility design of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Adaptive Staged SBRT)
Number analyzed (Participants) | 15
Participants
  met primary endpoint of CDD >3 mm | 1
  did not meet primary endpoint of CDD >3 mm | 14

2. Primary Outcome: Number of Participants Demonstrating Successful Radiographic Response of the Spinal Tumor
Description: Successful radiographic response of the spinal tumor was determined by achieving of a 10% reduction in epidural volume or thecal sac compression (i.e., ~10% absolute increase in thecal sac patency (TSP)) following treatment, on either of their MRI imaging or CT myelogram scans. Data was summarized using standard descriptive statistics; formal hypothesis testing was not performed. Confidence intervals for the true proportion using Clopper-Pearson exact confidence interval were not conducted. Since this is a feasibility study no power calculation was done.
Time Frame: Up to 10 weeks after first treatment
Population: Data was not collected and analyzed for 10 participants due to no post-treatment MRI or CT myelograms being obtained. Imaging was unable to be conducted for these 10 participants due to either a decline in subjects' clinical status or death. Confidence intervals were not determined given data limitations and had no impact due to feasibility design of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Adaptive Staged SBRT)
Number analyzed (Participants) | 14
Participants
  Participants with significant TSP difference | 8
  Participants without significant TSP difference | 6

3. Secondary Outcome: Change in Ambulation (Mobility)
Description: Ambulation was assessed as a functional outcome by the treating physician. Scoring was adapted from the ICORG Phase III trial, ASTRO 2014. Mobility scores were assigned as follows: 1 = ambulatory without aid; 2 = ambulatory with aid; 3 = not ambulatory; and 4 = paraplegia. Basic descriptive statistics were used to assess changes in ambulation from baseline.
Time Frame: 10 weeks after first treatment
Measure: Mean (Standard Deviation); unit: Change in ambulation measure score
Arm/Group | Treatment (Adaptive Staged SBRT)
Number analyzed (Participants) | 24
Change in ambulation measure score | .3 (3)

4. Secondary Outcome: Change in Pain Control in Terms of Pain Scores as Measured by the Numeric Pain Rating Scale (NPRS) Estimation
Description: Participants were asked to provide a numeric value using the NPRS to describe their pain intensity. The NPRS is a unidimensional assessment tool which measures pain on an 11-point (0-10) numeric scale where "0" represents no pain and "10" represents extreme pain. Higher scores are indicative of worsening pain intensity.
Time Frame: Up to 10 weeks after first treatment
Population: Data was not collected and analyzed for all patient due to diminishing clinical status or death.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (Adaptive Staged SBRT)
Number analyzed (Participants) | 22
score on a scale
  pretreatment best | 4.3 (3)
  pretreatment worst | 7.18 (2.8)
  weeks 2-4 best: number analyzed (Participants) | 14
  weeks 2-4 best | 3.46 (2.6)
  weeks 2-4 worst: number analyzed (Participants) | 14
  weeks 2-4 worst | 5.85 (3.7)
  weeks 8-10 best: number analyzed (Participants) | 7
  weeks 8-10 best | 2.85 (3.6)
  weeks 8-10 worst: number analyzed (Participants) | 7
  weeks 8-10 worst | 6 (3.5)

5. Secondary Outcome: Health Related Quality of Life Scores (FACT-G)
Description: Health-related Quality of Life was measured using Functional Assessment of Cancer Therapy - General (FACT-G) a 27-item questionnaire designed to measure four domains of Quality of Life in cancer patients assessed over the previous 7-day period: physical well-being (7 questions), social/family well-being (7 questions), emotional being (6 questions), and functional well-being (7 questions). Participant responses are assessed using a 5 point Likert-type scale ranging from 0 (Not at all) to 4 (Very much). A FACT-G total score is computed as the sum of the four subscale scores, provided the overall item response is at least 80% (i.e. at least 22 of the 27 items answered) and has a possible range of 0-108 points. Negatively worded items are reverse scored prior to summing so that higher subscale and total scores indicate a better overall health state corresponding Quality of Life.
Time Frame: Up to 3 months following first treatment
Population: Data was not collected and analyzed for 15 participants due to either a decline in subjects' clinical status or death.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (Adaptive Staged SBRT)
Number analyzed (Participants) | 9
score on a scale | 5 (3)

6. Secondary Outcome: Incidence of Any Grade Greater Than or Equal to 3 Treatment-related Toxicity, Scored Using CTCAE, v. 4
Description: Data will be reported in a descriptive manner to describe any incidence of greater than or equal to 3 treatment related toxicity
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Adaptive Staged SBRT)
Number analyzed (Participants) | 24
Participants | 0

7. Secondary Outcome: Incidence of Grade Greater Than or Equal to 2 Radiation-induced Lung Toxicity (CTCAE), Version (v.) 4
Description: Data will be reported in a descriptive manner to describe any incidence of grade 2 or greater related radiation induced lung toxicity
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Adaptive Staged SBRT)
Number analyzed (Participants) | 24
Participants | 0

8. Secondary Outcome: Overall Survival
Description: Data will be reported in a descriptive manner.
Time Frame: From study registration to death, censored at the date of data collection, assessed up to 2 years
Population: patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Adaptive Staged SBRT)
Number analyzed (Participants) | 13
Participants | 13

9. Secondary Outcome: Progression-free Survival
Description: Data will be reported in a descriptive manner.
Time Frame: From study registration to date of disease progression or death, censored at the date of data collection, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Adaptive Staged SBRT)
Number analyzed (Participants) | 13
Participants | 12

ADVERSE EVENTS:
Time Frame: Up to time of final imaging visit, approximately 8-10 weeks following initial treatment, unless otherwise clinically indicated
Arm/Group | Treatment (Adaptive Staged SBRT)
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 5/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Adaptive Staged SBRT) (N=24)
Fatigue (General disorders) | 5
Urinary Frequency (Increased) (Renal and urinary disorders) | 1 — Grade 1. Related to Sunitinib
Esophagitis (Gastrointestinal disorders) | 1 — Grade 2
Dysphagia (Gastrointestinal disorders) | 1 — Grade 2
Diarrhea (Gastrointestinal disorders) | 1 — Grade 3. Related to Afatinib treatment
Anorexia (Metabolism and nutrition disorders) | 1 — Grade 3. Related to Afatinib treatment
Mucositis oral (Gastrointestinal disorders) | 1 — Grade 3
Conjuctivitis (Eye disorders) | 1 — Grade 2
Paronychia (Infections and infestations) | 1 — Grade 2
Nausea (Gastrointestinal disorders) | 1 — Grade 2
Weight Loss (Investigations) | 1 — Grade 2
Rash (nonspecific) (Skin and subcutaneous tissue disorders) | 1 — Grade 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 — Grade 2
Urinary Tract Infection (Infections and infestations) | 1 — Grade 3
Anemia (Blood and lymphatic system disorders) | 1 — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT02527304/Prot_SAP_000.pdf